CLINICAL TRIAL: NCT04481308
Title: Reliability of Non-invasive Carbon Dioxide Monitoring During Conscious Sedation for Adult Endoscopic Retrograde Cholangiopancreatography Patients
Brief Title: Non-invasive Carbon Dioxide Monitoring and Endoscopic Retrograde Cholangiopancreatography Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Fouad Yones, Resident of anesthesia and intensive care, Assiut University
Other Study IDs: non-invasive co2 monitoring
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Patient Monitoring
Keywords: Non-Invasive; CO2 Monitoring; Conscious Sedation; Adult ERCP
MeSH Terms: interventions — Propofol; Fentanyl

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: propofol (2 mg/kg) and fentanyl (1ug/kg) and 4 liters O2 flow through nasal cannula — propofol (2 mg/kg) and fentanyl (1ug/kg) and 4 liters O2 flow through nasal cannula

SUMMARY:
CO2 monitoring through non-invasive methods to provide an early warning of hypoventilation during procedural sedation.

DETAILED DESCRIPTION:
Many patients become hypoxic during endoscopic retrograde cholangiopancreatography (ERCP). Following induced sedation, hypoxia or hypercapnia may follow . Monitoring the CO2 level during respiration (capnography) is non-invasive, easy to do, relatively inexpensive, and has been studied extensively . End-tidal carbon dioxide is the level of CO2 released at the end of an exhaled breath . Capnography provides information about ventilation, perfusion and metabolism . Capnography devices are configured as either side stream or mainstream. Side stream devices can monitor both intubated and non-intubated patients, while mainstream devices are most often limited to intubated patients .

The Dual guard (made in China) sets a standard in endoscopic practices; it incorporates an endoscopy bite block with oxygen delivery and CO2 monitoring for use in upper endoscopy procedures through to recovery . It improves patient safety and meets current guidelines for consciously sedated patients. The Comfort Rest Bite Block fits securely in the mouth, protecting both endoscope and patients' teeth. Simultaneous oral and nasal O2 delivery and CO2 sampling for patients undergoing upper GI endoscopy, in either a lateral or supine position. Arterial blood gas test results show the patient's acid-base balance, which is measured by the hydrogen ion concentration present in the blood, its oxygen saturation, partial pressure of oxygen (PaO2), partial pressure of carbon dioxide (PaCO2), concentration of bicarbonate (HCO3), base excess and base deficit . Itcan provide information about a surgical patient's physiological state, oxygenation, ventilation and indicate the primary source of a disturbance (ie, respiratory or metabolic) in homeostasis .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-50 years.
* Males or females.
* Elective Endoscopic Retrograde Cholangiopancreatography Patients

Exclusion Criteria:

* Patient with abnormal renal function test.
* Patient with history of chronic chest disease like asthma or Chronic obstructed pulmonary diseases.
* Patients with a history of systemic illness like hypertension and diabetes.
* Cardiac patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients aged 20-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
mparison between CO2 measurement from non-invasive method (Dual guard) during conscious sedation for ERCP and invasive method (arterial blood gases). | october 2020
  mparison between CO2 measurement from non-invasive method (Dual guard) during conscious sedation for ERCP and invasive method (arterial blood gases).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Medicin, Asyut
  - Samar, Asyut